CLINICAL TRIAL: NCT06329674
Title: Evaluate the Efficacy and Safety of the Combination of A51R3 and AJU-A51 Compared With the Combination of A51R3 and A51R2 in Patients With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of AJU-A51 in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AJU Pharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20DM30203
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AJU-A51+A51R2 placebo+A51R3 (Experimental)
  Interventions: Drug: AJU-A51; Drug: A51R3; Drug: A51R2 Placebo
- AJU-A51 placebo+A51R2+A51R3 (Experimental)
  Interventions: Drug: A51R2; Drug: A51R3; Drug: AJU-A51 Placebo

INTERVENTIONS:
Drug: AJU-A51 — Subjects take the investigational products once a day for 24 weeks.
  Arms: AJU-A51+A51R2 placebo+A51R3
Drug: A51R2 — Subjects take the investigational products once a day for 24 weeks.
  Arms: AJU-A51 placebo+A51R2+A51R3
Drug: A51R3 — Subjects take the investigational products once a day for 24 weeks.
Drug: AJU-A51 Placebo — Subjects take the investigational products once a day for 24 weeks.
  Arms: AJU-A51 placebo+A51R2+A51R3
Drug: A51R2 Placebo — Subjects take the investigational products once a day for 24 weeks.
  Arms: AJU-A51+A51R2 placebo+A51R3

SUMMARY:
A multicenter, randomized, double-blind, parallel group, placebo-controlled, phase 3 study to evaluate the efficacy and safety of the combination of A51R3 and AJU-A51 compared with the combination of A51R3 and A51R2 in patients with Type 2 diabetes mellitus who have inadequate glycemic control with the combination of A51R3 and A51R2

ELIGIBILITY:
Inclusion Criteria:

* Those who voluntarily signed the informed consent to participate in this study.
* Adults aged 19-75 years.
* Those diagnosed with type 2 diabetes mellitus.
* 7% ≤ HbA1c ≤ 10.5%
* FPG ≤ 270 mg/dL
* BMI ≤ 40 kg/㎡
* Subjects able to understand the study, comply with study procedures, and attend all scheduled visits.

Exclusion Criteria:

* Those who suffered from acute or chronic metabolic acidosis, lactic acidosis and diabetic ketoacidosis.
* Those who had genetic disorders such as galactose intolerance, Lapp lactose deficiency, or glucose-galactose malabsorption.
* Those with heart failure (NYHA class II~IV) or who had suffered from heart failure.
* Those with a history of malignant tumor within 5 years
* Those who have a clinically significant liver disease
* Those who have a clinically significant renal disease
* SBP > 180 mmHg or DBP > 110 mmHg
* Those who had allergic reaction to main ingredients or components of the investigational products.
* Patients planning to become pregnant or of childbearing potential, but not using any recognized contraceptive method
* Females who are pregnant or breastfeeding.
* AST or ALT ≥ LRN*3
* TG ≥ 500 mg/dL

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Changes in HbA1c | 24th week
  Changes in HbA1c at the 24th week after the administration of investigational products from the baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong JH, Kim MJ, Min KW, Won JC, Kim TN, Lee BW, Kang JG, Kim JH, Park JH, Ku BJ, Lee CB, Kim SY, Shon HS, Lee WJ, Park JY. Efficacy and safety of a fixed-dose combination of dapagliflozin and linagliptin (AJU-A51) in patients with type 2 diabetes mellitus: A multicentre, randomized, double-blind, parallel-group, placebo-controlled phase III study. Diabetes Obes Metab. 2025 Jan;27(1):81-91. doi: 10.1111/dom.15985. Epub 2024 Oct 7. PMID 39375869